CLINICAL TRIAL: NCT03676959
Title: An Open-label, Dose-escalation, Bi-weekly Phase I Clinical Trial in Treating Patients With Recurrent or Metastatic Cervical Cancer
Brief Title: A Clinical Study of PD-L1 Antibody ZKAB001（Drug Code） in Recurrent or Metastatic Cervical Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NTL-LEES-2017-02
Record Dates: First submitted 2018-09-12; First posted 2018-09-19 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZKAB001 5mg/kg (Experimental): Three or six patients will be treated with the dose of 5 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 5mg/kg
- ZKAB001 10 mg/kg (Experimental): Three or six patients will be treated with the dose of 10 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 10mg/kg
- ZKAB001 15 mg/kg (Experimental): Three or six patients will be treated with the dose of 15 mg/kg/time of ZKAB001 IV bi-weekly. DLT will be observed within 28 days after administration.
  Interventions: Drug: ZKAB001 15mg/kg

INTERVENTIONS:
Drug: ZKAB001 5mg/kg — 5mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 5mg/kg
Drug: ZKAB001 10mg/kg — 10mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 10 mg/kg
Drug: ZKAB001 15mg/kg — 15mg/kg/times bi-week IV administration of ZKAB001
  Other Names: PD-L1 monoclonal antibody
  Arms: ZKAB001 15 mg/kg

SUMMARY:
This is a Phase 1, open-label, dose-escalation, and multidose study, aiming to investigate the safety, tolerability and pharmacokinetics(PK) of ZKAB001 (a fully human monoclonal antibody targeting the Programmed Death - Ligand 1 (PD-L1) membrane receptor on T lymphocytes and other cells of the immune system) administered every 14 days in subjects with recurrent or metastatic cervical cancer.

DETAILED DESCRIPTION:
The study will consist of 4 periods: Screening (up to 28 days), Lead-in period (Day -28), Treatment (up to 24 cycles or 1 year, whichever occurs first), and Follow-up (up to 1 year). There will be a lead-in period on Day -28 for each dose escalation cohort in which the single-dose pharmacokinetics of ZKAB001 will be characterized prior to initiation of continuous dosing in the first cycle of treatment. The lead-in period duration, PK time-points, doses and/or regimens used in subsequent cohorts may be modified based on the exposure (AUC) observed during the lead-in period (although the number of PK samples will not be increased). Treatment of continuous dosing is up to 24 cycles or 1 year, until as per investigator's opinion, subjects experience disease progression (evaluated by RECIST 1.1 and immune-related response criteria irRECIST), no clinical benefit, or intolerable toxicity. If investigators suspect subjects experience pseudoprogression or has evidence to prove "mixed response", subjects can continue to accept treatment as investigator decided.

The study was divided into two stages. After the recommended phase II dose (RP2D) is determined in the first stage, the sample size will be amplified with RP2D in the second stage. When a total of 15 cases are included in the two stages, an interim analysis will be conducted to decide whether to expand the total number of cases to 60 based on the results of the analysis. If more than 2 cases of response will be observed in 15 cervical cancer subjects, 45 cases (with a total sample size of 60 cases) could be included to further observe the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily gives written informed consent to participate in the study.
2. Female subjects aged≥18 years.
3. Recurrent or metastatic cervical cancer was diagnosed by histopathology or cytology and received first-line platinum-containing regimens that failed or could not be tolerated. The definition of first-line failure: progress during adjuvant therapy or within 6 months after the end of treatment, and the first progress after palliative treatment.
4. Based on RECIST1.1, imaging evaluation confirmed that there was at least one measurable disease.
5. Eastern Cooperative Oncology Group（ECOG） performance status of 0 or 1, with estimated life expectancy of at least 3 months.
6. Adequate blood routine, hepatic and renal function:

1) Absolute neutrophil count（ANC）≥109/L 2) Platelets ≥100x109/L 3) Hemoglobin ≥9g/dL 4) Serum albumin ≥2.8g/dL 5) Bilirubin ≤1.5x Upper limit of normal（ULN） 6) ALT and AST ≤1.5xULN, if If liver metastases are present, alanine transaminase（ALT） and aspartate transaminase（AST） should be ≤5xULN 7) Creatinine clearance rate ≥50ml/min (Cockcroft-Gault equation) 7.Female reproductive subjects should take effective contraception during the study period and within 3 months after the study treatment period. The serum or urine human chorionic gonadotropin （HCG）examination must be negative within 7 days before the subject is enrolled.

Exclusion Criteria:

1. There are known active or suspected autoimmune diseases. Those who are in a stable state and do not need systemic immunosuppressive therapy can be included.
2. Patients are using immunosuppressive agents, or systemic, or absorbable topical corticosteroid medications to achieve immunosuppressive purposes (doses >10mg/day prednisone or equivalent), which is ongoing 2 weeks before enrollment.
3. Have received any form of organ transplantation, including allogeneic stem cell transplantation.
4. Known allergy to macromolecular protein inhibitors or any of the components of ZKAB001.
5. Suffering from other malignant tumors other than this diseases in 5 years except for skin basal cell and squamous cell carcinoma.
6. Central nervous system metastases with clinical symptoms (such as cerebral edema and brain metastases requiring corticosteroid intervention). Previous treatment with brain or meningeal metastasis, such as clinical stabilization (MRI) less than 2 months, or systemic corticosteroid (dose >10mg/day prednisone or equivalent) less than 2 weeks.
7. Patients with clinical symptoms or diseases of the heart that cannot be well controlled, such as heart failure above New York Heart Association ( NYHA ) 2 grade, unstable angina pectoris, myocardial infarction in 1 year, and clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, have left ventricular ejection fraction < 50% at rest in the ultrasound cardiogram.
8. Patients who had received radiotherapy, chemotherapy, surgery or molecular targeted therapy before, were given less than 4 weeks.
9. Within 14 days before the first use of the drug, any active infection requiring systematic anti-infective treatment.
10. Human immunodeficiency virus (HIV) positive, untreated active hepatitis (hepatitis B surface antigen positive and peripheral blood HBV-DNA titer ≥ 500IU/ml or positive copy number detected by the research center; hepatitis C virus antibody positive)
11. There is a history of active pulmonary tuberculosis within 1 year before entering the group.
12. The patient is participating in other clinical studies or is less than 1 month away from the end of the previous clinical study.
13. Patients may need to receive other systemic cancer treatment during study period.
14. Received blood transfusion and hematopoietic stimulating factors, such as colony stimulating factor, erythropoietin, thrombopoietin, etc., within 14 days before screening.
15. Prior therapy with an anti-PD 1, anti-PD L1, or anti-CTLA-4 (Cytotoxic T lymphocyte Antigen-4) antibody (or any other agents that target immunoregulatory receptor).
16. Subjects who received live vaccine within 4 weeks before screening.
17. History of mental drug abuse, alcohol abuse or drug abuse.
18. Pregnant or lactating women.
19. Any mental condition that prevents the understanding or provision of an informed consent.
20. It is determined by the investigator that the patient has other factors that may lead to the termination of the study, such as other serious diseases or serious laboratory test abnormalities or other factors that may affect the safety of the patients, family or social factors that may affect the study data and sample collection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 101 (Estimated)
Dates: Start 2018-08-16 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
RP2D | 28 days after first dose
  Recommended phase II dose.
Objective response rate | 2 years
  The proportion of subjects who achieved the best objective response rate (PR or CR).
Tolerance | 2 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Effect of ZKAB001 on T cell function and cytokine expression | through study completion, an average of 2 years
  The response of CD4+ and CD8+ cells to tumor at baseline and after each administration will be detected by flow cytometry.
The number of subjects presenting detectable anti drug antibodies (ADAs) | through study completion, an average of 2 years
  To evaluated the number of subjects presenting detectable anti drug antibodies (ADAs).
Receptor occupancy | through study completion, an average of 2 years
  Monocytes will be isolated from peripheral blood before each cycle of administration, and the receptor occupancy of PD-L1 on CD3+T cells will be determined.
PD-L1 expression | through study completion, an average of 2 years
  Detection of PD-L1 expression in tumor tissues.
progression free survival（PFS） | through study completion, an average of 2 years
  Evaluate the PFS of the study population
overall survival | through study completion, an average of 2 years
  Evaluate the OS of the study population
duration of response | through study completion, an average of 2 years
  Evaluate the DOR of the study population
best of response | through study completion, an average of 2 years
  Evaluate the BOR of the study population

CONTACTS AND LOCATIONS:
Overall Officials: lingying Wu, M.D, Study Director — Tumor Hospital of the Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] An J, Tang J, Li BX, Xiong H, Qiu H, Luo L, Wang L, Wang D, Zhou Q, Xu Q, Song H, Zhang Y, Zhang H, Li Y, Yu X, Zhang J, Ng R, Zhao W, Wong M, Dai X, Li G, Wu L. Efficacy and Safety of the Anti-PD-L1 mAb Socazolimab for Recurrent or Metastatic Cervical Cancer: a Phase I Dose-Escalation and Expansion Study. Clin Cancer Res. 2022 Dec 1;28(23):5098-5106. doi: 10.1158/1078-0432.CCR-22-1280. PMID 36136294